CLINICAL TRIAL: NCT04385004
Title: Characterization of the Clinical, Biological and Histological Pulmonary and Renal Damage Associated With the SARS-CoV-2 Syndrome in Patients Admitted in the Intensive Care Unit
Brief Title: Clinical, Biological and Histological Pulmonary and Renal Damage Associated With the SARS-CoV-2 Syndrome in Patients Admitted in ICU
Acronym: PR-Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7815
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Covid-19; SARS-CoV-2; Inflammatory cytokine; Sepsis; ICU; Tbular necrosis; Ischemia; Pulmonary damage; Renal damage; Kidney damage
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Sepsis; Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Renal damage in patients hospitalized for ARDS in the ICU can also be related to multiple causes including, but not limited to, the consequences of hemodynamic fluctuations in these patients or the use of nephrotoxic drugs responsible for acute post-ischemic or toxic tubular necrosis. Frequently observed abnormalities of cioagumation may also have a potential impact on renal structures, particularly glomerular capillaries.

The researchers wish to characterize and phenotype the renal impairment of patients hospitalized in intensive care with tables of severe Covid19 infections in ARDS: clinical, biological and histological (by performing post-mortem biopsies).

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Diagnosed Covid-19 by RT PCR
* Hospitalized in intensive care for management of complications related to Covid-19 from March 1, 2020 to April 20, 2020
* Patient not having expressed his or her opposition, after information, to the re-use of his or her data for the purposes of this research.

Exclusion Criteria:

- Subject who expressed opposition to participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed Covid-19 by RT PCR
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Analysis of Clinical, Biological and Histological Pulmonary and Renal Impairment Related to SARS-CoV-2 | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service Reanimation Medicale, Strasbourg, France

REFERENCES:
- [Derived] Beloncle F, Studer A, Seegers V, Richard JC, Desprez C, Fage N, Merdji H, Pavlovsky B, Helms J, Cunat S, Mortaza S, Demiselle J, Brochard L, Mercat A, Meziani F. Longitudinal changes in compliance, oxygenation and ventilatory ratio in COVID-19 versus non-COVID-19 pulmonary acute respiratory distress syndrome. Crit Care. 2021 Jul 15;25(1):248. doi: 10.1186/s13054-021-03665-8. PMID 34266454